CLINICAL TRIAL: NCT05746741
Title: Telehealth Intervention Strategies for WIC (THIS-WIC)- Michigan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency); State of Michigan WIC Program (Unknown); RTI International (Other)
Responsible Party: Principal Investigator, Erin Hennessy, Assistant Professor, Division of Nutrition Interventions, Communication and Behavior Change Director ad interim, ChildObesity180 Friedman School of Nutrition Science and Policy, Tufts University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 202112-01-EA / STUDY00002536
Record Dates: First submitted 2023-02-16; First posted 2023-02-28 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Telehealth; Nutrition Education; Breast Feeding; Dietary Intake; WIC
Keywords: Telehealth; WIC; nutrition education; breast feeding; dietary intake
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Study participants will be clients at local WIC agency sites where either the telehealth solution is offered or where only usual care is available (control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth solution (Experimental): Telehealth solution offered
  Interventions: Behavioral: Telehealth solution
- Control (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Telehealth solution — Video conferencing
  Arms: Telehealth solution

SUMMARY:
With funding through the United States Department of Agriculture (USDA) and Tufts University's Telehealth Intervention Strategies for WIC (THIS-WIC), Michigan's (MI) WIC department will pilot telehealth opportunities as a means of delivering services to WIC Clients. This video conferencing pilot looks to improve and/or remove barriers. Implementing a pilot program in select local agencies to utilize technology would allow clients to connect with a WIC Registered Dietitian (RD) or an International Board-Certified Lactation Consultant (IBCLC). Videoconferencing could open new opportunities for leveraging the extensive expertise of the nutrition and lactation workforce in WIC agencies to address rural and remote locations and travel considerations.

The purpose of this study will be to evaluate the effectiveness of this telehealth solution.

DETAILED DESCRIPTION:
Michigan WIC Agency will pilot telehealth opportunities as a means of delivering services to WIC Clients.This video conferencing pilot looks to improve and/or remove barriers such as negative clinic experiences (long wait times or poor customer service), lost time from work (creating job risk and lost wages), inconvenient WIC clinic locations and appointment times, and lack of transportation. Implementing a pilot program in select local agencies to utilize technology would allow clients to connect with a WIC Registered Dietitian (RD) or an International Board-Certified Lactation Consultant (IBCLC). Videoconferencing could open new opportunities for leveraging the extensive expertise of the nutrition and lactation workforce in WIC agencies to address rural and remote locations and travel considerations. Additional urban locations, where clients lack transportation or use of public transportation presents a barrier to traveling to subsequent WIC appointments, will also be included in the pilot. Local agencies in rural and urban areas with similar caseloads will serve as controls to compare outcomes between offering telehealth and conducting IBCLC and RD appointments in person.

The purpose of this study is to evaluate the effectiveness of this telehealth solution by having clients complete surveys on their comfortability using telehealth and their satisfaction with the telehealth appointment. Additionally, secondary demographic and other nutrition-related information about study participants is already collected in the MIS and will be utilized.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Breastfeeding women
* postpartum women with children in the age range of 0 to 5 years

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Satisfaction with the telehealth solution | During the study period, approximately 18 months
  WIC clients satisfaction with nutrition education and breastfeeding support offered via the telehealth solution compared to usual care. Data will be collected, and this outcome measure will be assessed via survey completion by study participants.

SECONDARY OUTCOMES:
Breastfeeding duration | During the study period, approximately 18 months
  Duration of breastfeeding in clients offered the telehealth solution compared to usual care. Data will be collected, and this outcome measure will be assessed via survey completion by study participants.
Attendance at scheduled appointments | During the study period, approximately 18 months
  WIC clients attendance at appointments when offered the telehealth solution compared to usual care. Data will be collected, and this outcome measure will be assessed via survey completion by study participants.
Dietary intake | During the study period, approximately 18 months
  Impact of the telehealth solution compared to usual care on dietary intake. Data will be collected, and this outcome measure will be assessed via survey completion by study participants.
Attitudes to breastfeeding and nutrition education | During the study period, approximately 18 months
  Impact of the telehealth solution compared to usual care on WIC clients' attitudes to breastfeeding and nutrition education. Data will be collected, and this outcome measure will be assessed via survey completion by study participants.
Barriers encountered in obtaining nutrition education and breastfeeding support | During the study period, approximately 18 months
  Impact of the telehealth solution compared to usual care on barriers encountered by WIC clients in obtaining nutrition education and breastfeeding support. Data will be collected, and this outcome measure will be assessed via survey completion by study participants.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Hennessy, PhD, Principal Investigator — Tufts University
Locations (1):
- Tufts University, Boston, Massachusetts, United States

REFERENCES:
- See also: Tufts Telehealth Intervention Strategies for WIC (THIS-WIC) website — https://thiswic.nutrition.tufts.edu/